CLINICAL TRIAL: NCT05468554
Title: Evaluation of Metformin Effect on the Fertility of Women Treated With 131I for Thyroid Cancer
Acronym: METHYR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/ABM/01/00100
Record Dates: First submitted 2022-07-08; First posted 2022-07-21 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Metformin; Iodine-131

STUDY DESIGN:
Intervention Model Description: Arm A - patients qualified to receive metformin and 131I treatment, arm B - patients receiving placebo and 131 I treatment. Arm C- observation group, patients undergoing thyroidectomy, characterized by low risk of disease progression, in this case, not qualified for the 131I treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind / placebo controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin (Experimental): patients qualified to receive metformin and 131I treatment
  Interventions: Drug: metformin; Radiation: Radioactive iodine (I-131)
- Placebo (Active Comparator): patients receiving placebo and 131 I treatment
  Interventions: Radiation: Radioactive iodine (I-131)
- Observational (No Intervention): observation group, patients after thyroidectomy, characterized by low risk of cancer progression, in this case, not qualified for 131I treatment

INTERVENTIONS:
Drug: metformin — Metformin will be used 3 times a day (3x500mg), starting in the first week with 1x1 tablet (1x500 mg for breakfast), in the second week, 2x1 tablet (500 mg for breakfast and 500 mg for dinner), from the 3rd week 3x1 tablet. (3x500mg with main meals). A gradual escalation of the dose is planned to the point of developing drug intolerance or toxicity that is unacceptable to the patient.
  Arms: Metformin
Radiation: Radioactive iodine (I-131) — Patients qualified to receive 131I treatment
  Arms: Metformin; Placebo

SUMMARY:
This study is aimed to investigate the metformin effect on the fertility of women treated with 131 I for thyroid cancer

DETAILED DESCRIPTION:
One of the most common types of endocrine cancer, especially in young women, is thyroid cancer. More than 90% of all thyroid cancers are differentiated thyroid cancers (DTC), including papillary thyroid cancer (PTC) and follicular cancer. Papillary thyroid cancer is considered as indolent tumour as progression free survival is 10 years of 98%. As per current knowledge and basing on current literature most of the PTC are considered to be low incidence of recurrence or metastasis, however, there are more invasive/aggressive types with very specific pathological and molecular characteristics. The aggressive variants of PTC were strictly associated with higher rates of extrathyroid extension, multifocality, and nodal and distant metastasis. Thyroidectomy followed by radioactive iodine 131 (131I) therapy, in higher stages of PTC disease to ablate residual thyroid cancer or treat metastases, significantly increase survival Metformin (1,1-dimethylbiguanide) is an oral antihyperglycemic drug. Orally administered metformin is absorbed into the blood in 40-60% of the drug dose. Maximum blood levels are reached after approximately 2.5 hours for the immediate-release formulation and 7 hours for the prolonged-release tablets. It is not metabolised in the liver, however, it is excreted unchanged by the kidneys, mainly through the renal tubules. Metformin is used in patients with type 2 diabetes and prediabetes as well as in insulin resistant state and in women with polycystic ovary syndrome (PCOS). Metformin works by lowering level of glucose in the blood by lowering its production by the liver and increasing the sensitivity to insulin by muscle and fat tissue. It also has a beneficial effect on serum lipids by reducing the concentration of triglycerides, total cholesterol, LDL-cholesterol and VLDL. Additionally, this drug has also several other biological effects such as anti-inflammatory, anticancer, hepatoprotective, cardioprotective, otoprotective, radioprotective and radio-sensitising.

Currently there is also a large evidential material for effectiveness of metformin therapy in re-establishing of reproductive functions and fertility in women with polycystic ovary syndrome.

Having proved the metformin restore of ovulation in PCOS and has antioxidant properties there are indications that metformin can be a therapy which will helps to maintain ovary follicle number on acceptable level. At present, there are no performed studies concerned on the evaluation of the potential beneficial effect of metformin application impact on fertility parameters in the group of women treated with 131I. Therefore, the proposed study will assess the effect of metformin intervention on the indirect parameters of fertility of women treated with 131I for papillary thyroid cancer

ELIGIBILITY:
Inclusion Criteria:

* Female subjects in reproductive age >18 <45.
* Subjects with diagnosed papillary thyroid carcinoma with various pathological, stage TNM (I-II).
* Subjects not treated with 131I.
* Serum TSH concentration 0.1-4.9 mU/l.
* Willingness to comply with protocol procedures.

Exclusion Criteria:

* Hypersensitivity to metformin.
* Subjects with polycystic ovarian syndrome or other diseases of the ovaries (primary / secondary ovarian failure).
* Subjects taking metformin during last week.
* Subjects with liver malfunction and abnormal hepatitis marker results (ALT and AST activity >3ULN.
* Subjects with eGFR below 45ml/min/1.73m2.
* Subjects with lactic acidosis or having history of metabolic acidosis.
* Subjects with serum AMH concentration below lower range norm.
* Subjects with history of congestive heart disease NYHA stage III/IV.
* Subjects with acute myocardial ischemia (CCS 3-4).
* Subjects with history of sepsis or severe infection.
* Subject with lung disease (uncontrolled asthma based on GINA 2000 Guidelines and COPD GOLD ≥ 3 stage).
* Positive result of pregnancy test or pregnancy planned during the study.
* Alcohol or other substance dependent syndromes.
* BMI <18.5 kg/m2.
* Accompanying diseases with poor prognosis in the opinion of the researcher.
* As per Investigator (or his designee) judgement, subject cannot participate in the study due to reasons (i.e. medical, psychiatric and/or social reason).
* Unreliability or lack of cooperation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in AMH, Inhibin B and FSH levels due to the action of metformin | 4 years
  The primary endpoint will be to evaluate the effect of metformin on the difference in serum AMH, inhibin B and FSH concentration and the number of antral follicles, assessed in the study groups consisted of the women with papillary thyroid cancer, treated with 131I, comparing received results during the randomized, V3, V4, V5 and V6 visits

SECONDARY OUTCOMES:
Assessment of the effect of metformin on the parameters of oxidative stress | 4 years
  To evaluate the metformin modulating impact on the concentrations of selected parameters of oxidative stress assessed in the study groups consisted of the women with papillary thyroid cancer, treated with 131I, comparing received results during the randomized, V3, V4, V5 and V6 visits
The evaluate of difference in serum concentration of selected parameters of apoptosis | 4 years
  To evaluate the effect of metformin on the difference in serum concentration of selected parameters of apoptosis between the study groups in women with papillary thyroid cancer, treated with 131I, comparing received results during the randomized, V3, V4, V5 and V6 visits
The evaluate of difference in expression in selected microRNA | 4 years
  To evaluate the effect of metformin on the difference of expression in selected microRNA between the study groups in women with papillary thyroid cancer, treated with 131I, between the randomized visit and V3, V4, V5 and V6 visit

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Adamska, Assoc.Prof., Principal Investigator — Medical University of Bialystok
Locations (1):
- Department of Endocrinology, Diabetology and Internal Medicine, Medical Univeristy of Bialystok, Bialystok, Poland